CLINICAL TRIAL: NCT06492174
Title: AGENT IDE: A Prospective, Randomized (2:1), Multicenter Trial to Assess the Safety and Effectiveness of the AgentTM Paclitaxel Coated PTCA Balloon Catheter for the Treatment of Subjects With In-Stent Restenosis (ISR)
Brief Title: A Clinical Trial to Assess the Agent Paclitaxel Coated PTCA Balloon Catheter for the Treatment of Subjects With In-Stent Restenosis (ISR) - Long Lesion Cohort
Acronym: AGENT IDE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 92294616
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: In-Stent Restenosis
Keywords: Drug coated balloon

STUDY DESIGN:
Intervention Model Description: A non-randomized, single arm cohort of subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- AGENT DCB 40 mm (Experimental): Agent DCB 40 mm is a Monorail Percutaneous Transluminal Coronary Angioplasty (PTCA) balloon catheter with a semi-compliant balloon coated with a formulation of paclitaxel (drug) and an excipient, Acetyl-Tri-n-butyl citrate (ATBC). The balloon catheter platform is based on the commercially available BSC Emerge™ PTCA balloon catheter system (K130391).
  Interventions: Device: AGENT DCB 40 mm

INTERVENTIONS:
Device: AGENT DCB 40 mm — Drug coated PTCA balloon catheter 40 mm size

SUMMARY:
The purpose of the AGENT IDE study is to assess the safety and effectiveness of the Agent Paclitaxel Coated PTCA Balloon Catheter in patients with in-stent restenosis (ISR) of a previously treated lesion of up to 36 mm in length (by visual estimate) in a native coronary artery 2.0 mm to 4.0 mm in diameter.

DETAILED DESCRIPTION:
Please see NCT04647253 for the prospective, randomized, multi-center, single blind trial comparing AGENT DCB to balloon angioplasty (POBA).

The Long Lesion Cohort is a non-randomized, single arm cohort of subjects with ISR of a previously treated lesion ≥ 26 mm and ≤ 36 mm in length (by visual estimate) in a native coronary artery 2.0 mm to 4.0 mm in diameter.

ELIGIBILITY:
Clinical Inclusion Criteria:

* Subject must be at least 18 years of age
* Subject (or legal guardian) understands the trial requirements and the treatment procedures, and provides written informed consent before any trial-specific tests or procedures are performed
* Subject is eligible for percutaneous coronary intervention (PCI)
* Subject is willing to comply with all protocol-required follow-up evaluation
* Women of child-bearing potential must agree to use a reliable method of contraception from the time of screening through 12 months after the index procedure

Angiographic Inclusion Criteria (visual estimate)

* In-stent restenosis in a lesion previously treated with either a drug-eluting stent or bare metal stent, located in a native coronary artery with a visually estimated reference vessel diameter (RVD) > 2.0 mm and ≤ 4.0 mm.
* Target lesion length must be ≤ 36 mm (by visual estimate) and must be covered by only one balloon.
* Target lesion must have visually estimated stenosis > 50% and < 100% in symptomatic patients (>70% and <100% in asymptomatic patients) prior to lesion pre-dilation.
* Target lesion must be successfully pre-dilated.

Note: Successful predilation/pretreatment refers to dilation with a balloon catheter of appropriate length and diameter, or pretreatment with directional or rotational coronary atherectomy, laser or cutting/scoring balloon with no greater than 50% residual stenosis and no dissection greater than National Heart, Lung, Blood Institute (NHLBI) type C. Thrombolysis in Myocardial Infarction (TIMI) grade flow in the target lesion must be >2

* If a non-target lesion is treated, it must be treated first and must be deemed a success.

Note: Successful treatment of a non-target lesion is defined as a residual stenosis of ≤ 30% in 2 near-orthogonal projections with TIMI 3 flow, as visually assessed by the physician, without the occurrence of prolonged chest pain or ECG changes consistent with MI.

Clinical Exclusion Criteria:

* Subject has other serious medical illness (e.g. cancer, congestive heart failure) that may reduce life expectancy to less than 24 months.
* Subject has current problems with substance abuse (e.g. alcohol, cocaine, heroin, etc.).
* Subject has planned procedure that may cause non-compliance with the protocol or confound data interpretation.
* Subject is participating in another investigational drug or device clinical study that has not reached its primary endpoint.
* Subject intends to participate in another investigational drug or device clinical study within 12 months after the index procedure.
* Woman who is pregnant or nursing. (A pregnancy test must be performed within 7 days prior to the index procedure, except for women who definitely do not have child-bearing potential.)
* Left ventricular ejection fraction known to be < 25%.
* Subject had PCI or other coronary interventions within the last 30 days.
* Planned PCI or CABG after the index procedure.
* STEMI or QWMI <72h prior to the index procedure.
* Cardiogenic shock (SBP < 80 mmHg requiring inotropes, IABP or fluid support).
* Known allergies against paclitaxel or other components of the used medical devices.
* Known hypersensitivity or contraindication for contrast dye that in the opinion of the investigator cannot be adequately pre- medicated.
* Intolerance to antiplatelet drugs, anticoagulants required for procedure.
* Platelet count < 100k/mm3 (risk of bleeding) or > 700k/mm3.
* Subject with renal insufficiency (creatinine ≥2.0 mg/dl) or failure (dialysis dependent).
* Subject has suspected or proven COVID-19 at present or within the past 4 weeks with resolution of symptoms.

Angiographic Exclusion Criteria (visual estimate)

* Target lesion is located within a bifurcation with planned treatment of side branch vessel.
* Target lesion is located within a saphenous vein or arterial graft.
* Thrombus present in the target vessel
* > 50% stenosis of an additional lesion proximal or clinically significant distal (>2.0mm RVD) to the target lesion.
* Patient with unprotected left main coronary artery disease. (>50% diameter stenosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2025-12-19 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Target Lesion Failure | 12-month
  The primary endpoint is the 12-month Target Lesion Failure (TLF) rate, defined as any ischemia-driven revascularization of the target lesion (TLR), myocardial infarction (MI, Q-wave and non-Q-wave) related to the target vessel, or cardiac death

CONTACTS AND LOCATIONS:
Overall Officials: Robert Yeh, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (11):
- United States (11):
  - Carondelet Medical Group St. Mary's Hospital, Tucson, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - Emory University Hospital, Atlanta, Georgia
  - Henry Ford Hospital, Detroit, Michigan
  - Columbia University Medical Center, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Lindner Center for Research and Education at Christ Hospital, Cincinnati, Ohio
  - UPMC Pinnacle Health, Wormleysburg, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Centennial Medical Center, Nashville, Tennessee
  - Baylor Heart and Vascular Hospital, Dallas, Texas